CLINICAL TRIAL: NCT03561480
Title: Effect of Postoperative Ferric Carboxymaltose After Simultaneous Bilateral Total Knee Arthroplasty : A Randomized, Controlled, Double-Blind Trial
Brief Title: Effect of Postoperative Ferric Carboxymaltose
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ferric Carboxymaltose 2
Record Dates: First submitted 2018-06-04; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Anemia; Knee Osteoarthritis; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric carboxymaltose group (Experimental): Ferinject®to be administered as IV drip infusion or undiluted bolus injection to consented patients with postoperative anemia after total knee arthroplasty.
  Interventions: Drug: Ferric carboxymaltose
- Placebo group (Active Comparator): Placebo(0.9% Normal Saline) to be administered as IV drip infusion or bolus injection to consented patients with postoperative anemia after total knee arthroplasty.
  Interventions: Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: Ferric carboxymaltose — Ferinject®to be administered as IV drip infusion or undiluted bolus injection with a minimum administration time of 15minutes (for 1000mg single administration) for body weight ≥50 Kg or 6 minutes (for 500mg single administration) for body weight <50Kg .
  Other Names: Ferinject®
  Arms: Ferric carboxymaltose group
Drug: 0.9% Normal Saline — Placebo will be in the form of normal saline administered over same time period as equivalent Ferinject® administration. IV drip infusion or undiluted bolus injection with a minimum administration time of 15 minutes (200mL as infusion or 20mL as bolus injection) for body weight ≥50 Kg or 6 minutes (100mL normal as infusion or 10mL as bolus injection) for body weight <50 Kg.
  Arms: Placebo group

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of postoperative intravenous ferric carboxymaltose in patients with anemia undergoing Simultaneous Bilateral Total knee replacement in terms of Quality of life (QOL) and objective measures (Hemoglobin and Iron parameters).

DETAILED DESCRIPTION:
Both preoperative and postoperative anaemia are common in patients undergoing total knee arthroplasty. Allogeneic RBC (red blood cell) transfusion and anaemia are related with higher postoperative mortality and morbidity. It is important to have a strategy of patient blood management.

Hb(hemoglobin) level of 10 g/dl will be used as a cut-off value for our study. In postoperative period in total knee arthroplasty for osteoarthritis, consented patients with postoperative anemia will be administered Ferinject® or placebo (normal saline) based on the results of randomization.

Study Group: Ferinject® administration as IV drip infusion or undiluted bolus injection with a minimum administration time of 15minutes (for 1000mg(milligram) single administration) for body weight ≥50 Kg (kilogram) or 6 minutes (for 500mg(milligram) single administration) for body weight < 50Kg( kilogram) .

Control Group: Placebo in the form of normal saline administration as same time period as equivalent Ferinject® administration. IV drip infusion or undiluted bolus injection with a minimum administration time of 15 minutes (200mL(milliliter) as infusion or 20mL(milliliter) as bolus injection) for body weight ≥50 Kg ( kilogram) or 6 minutes (100mL normal as infusion or 10mL(milliliter) as bolus injection) for body weight <50 Kg (kilogram).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age and signed written informed consent
* Patients scheduled to undergo major orthopaedic surgery (hip or knee arthroplasty or back surgery)
* Hb < 10.0 g/dl after operation
* Ferritin < 100 μg/l or 100-300 with transferrin saturation < 20%

Exclusion Criteria:

* Suspicion of iron overload (Ferritin >300 μg/l or/and transferrin saturation>50%)
* Active severe infection/inflammation (defined as serum C reactive protein > 20 mg/l) or diagnosed malignancy
* Folate-and/or Vitamin B12 deficiency (according to local lab reference range)
* Known history of hepatitis B/C or HIV-positive
* Liver values 3 times higher than normal
* Immunosuppressive or myelosuppressive therapy
* A concurrent medical condition(s) that, in the view of the investigator, would prevent compliance or participation or jeopardize the health of the patients.
* Pregnancy or lactation
* Transfusion within 1 month prior to study inclusion, erythropoietin treatment with in the last 4 weeks, any iron treatment within 4 weeks prior to the inclusion in the trail
* Participation in any other therapeutic trial within the previous month
* History of thromboembolic events in the family or the patient
* Severe peripheral, coronary or carotid artery disease
* Bodyweight < 50 kg
* Patients not able to understand the German language

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-11 (Estimated); Primary Completion 2019-06-11 (Estimated); Study Completion 2019-12-11 (Estimated)

PRIMARY OUTCOMES:
Hb increase from baseline till day of surgery | Postoperative 8 weeks from baseline
  Hb increase from baseline till day of surgery

SECONDARY OUTCOMES:
Percentage of patients requiring alternative anaemia management therapy | Percentage of patients requiring alternative anaemia management therapy up to 8weeks
  Percentage of patients requiring alternative anaemia management therapy
Self-reported patient assessment of EQ-5D (EuroQol-5 dimension ) | baseline and postoperative 4, 8 weeks
  Self-reported patient assessment of EQ-5D (EuroQol-5 dimension )
WOMAC(Western Ontario and McMaster University Arthritis Index ) scale | baseline and postoperative 2, 4, 8 weeks
  WOMAC(Western Ontario and McMaster University Arthritis Index ) scale
Brief pain inventory | baseline and postoperative 2, 4, 8 weeks
  Brief pain inventory

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Study Chair — The Catholic Univerisity of Korea Seoul St Mary's hospital

IPD SHARING:
Plan to Share IPD: Undecided